CLINICAL TRIAL: NCT07031674
Title: Comparing Efficacy and Safety of Telitacicept and Belimumab in Lupus Nephritis: A Retrospective Multicenter Cohort Study.
Status: Completed | Type: Observational
Sponsor: Yipeng Liu (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor-Investigator, Yipeng Liu, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2025(102)
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-07

CONDITIONS: Lupus Nephritis; Belimumab
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Telitacicept group: The participants in the study had previously used telitacicept as a therapeutic drug.
- The Belimumab group: The participants in the study had previously used belimumab as a therapeutic drug.

SUMMARY:
The objective of this observational study is to compare the efficacy and safety of telitacicept and belimumab in the treatment of lupus nephritis in patients aged 18-65 years with lupus nephritis. The main question it aims to answer is: What are the response rates of the two drugs for the main renal therapy in the lupus nephritis population? Which drug has better efficacy and safety? This study is a retrospective study. The participants will not receive any treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 65 years old;
* Meets the revised SLE classification criteria of the American College of Rheumatology in 1997 or the SLE diagnostic classification criteria issued by EULAR/ACR in 2019;
* Urine protein quantification ≥ 1g/d, or urine PCR ≥ 1g/g, or qualitative urine protein test in urine routine ≥ 1+;
* Patients who have been using telitacicept or belimumab for at least 12 weeks.

Exclusion Criteria:

* Having active central nervous system diseases;
* eGFR < 30 mL/min/1.73m², or undergoing hemodialysis or kidney transplantation;
* Pregnant women, or those who are about to become pregnant in the near future, or lactating women;
* Participants who are simultaneously participating in other clinical studies;
* Patients who have received telitacicept or belimumab treatment for less than 12 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion period is from March 1, 2021 to March 1, 2024. Patients who visited the First Affiliated Hospital of Shandong University Medical University, the Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Wuhan University People's Hospital, and the Department of Nephrology of Capital Medical University Affiliated Beijing Friendship Hospital for clinical diagnosis of lupus nephritis were included.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
The response rate for major kidney treatments | From baseline to the end of 1-year treatment period
  1. 24-hour urine PCR ≤ 0.7 g/g (70 mg/mmol);
  2. eGFR decline does not exceed 20% of the baseline or is ≥ 60 ml/min/1.73 m2;
  3. No rescue treatment was adopted due to treatment failure.

SECONDARY OUTCOMES:
Complete renal response rate | From baseline to the end of 1-year treatment period
  1. 24-hour urine PCR < 0.5 g/g (50 mg/mmol);
  2. Renal function is stable or has improved (by no more than 10%-15% compared to the baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No